CLINICAL TRIAL: NCT05931614
Title: Unlimited or Restricted Fluid Intake in Patients with Heart Failure: a Non-inferiority Randomized Controlled Trial
Brief Title: Unlimited or Restricted Fluid Intake in Patients with Heart Failure
Acronym: FLUID-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Collaborators: Capio Sankt Görans Hospital (Other); Ersta Hospital, Sweden (Other)
Responsible Party: Principal Investigator, Carolin Nymark, Director of Nursing Development, Region Stockholm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K 2023-3124
Record Dates: First submitted 2023-06-16; First posted 2023-07-05 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
Keywords: Quality of life; Intervention; Thirst distress; Symptoms; Physical capacity; Hospital readmissions; Lung ultrasound; Fluid intake; B-lines; NT-ProBNP; Heart failure; Fluid restriction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Free fluid intake (Experimental): Patients have no restrictions of fluid intake
  Interventions: Behavioral: Free fluid intake
- Restricted fluid intake (No Intervention): Patients are recommended a restricted fluid intake of 1500 mL/day

INTERVENTIONS:
Behavioral: Free fluid intake — Patients are recommended a free fluid intake
  Arms: Free fluid intake

SUMMARY:
Heart failure is the most common cause of admission to hospital and is associated with high morbidity and mortality. Treatment options consist of medical- and device treatment and self-care strategies, where fluid restriction has been one of the components in the self-care management of patients with chronic heart failure. The medical treatment has progressed and improved over the years and considerably over the last few years, which has decreased symptoms and improved physical function of these patients. Despite our great success in the medical treatment of heart failure, we still face challenges in hospital readmissions and treatment strategies. It contributes to the increased need of evidence on, if and how, fluid intake and fluid restriction should be used as a self-care method. Fluid restriction as a self-care treatment is still commonly recommended in heart failure management although the scientific clinical evidence is lacking. Fluid restriction is associated with a higher degree of thirst and lower rated quality of life, and there is no consensus on how fluid restriction should be used, no plan for individualized treatment and no agreement on how fluid restriction should be a part of the patient self-care treatment. There is therefore a need for knowledge on how heart failure patients are affected by fluid restriction regarding clincal signs and symptoms of heart failure, quality of life, physical function, readmission to hospital or heart failure events. The primary aim of the study is to investigate whether a free fluid intake is safe compared to a restricted fluid intake, regarding clinical signs of heart failure measured as the presence of B-lines and/or an increase in NT-proBNP. The secondary aim is to clarify whether an unlimited fluid intake can improve quality of life and reduce thirst without affecting heart failure symptoms, physical activity, hospital readmissions and/or heart failure events.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with left ventricual heart failure (HFrEF, HFmEF)
* Physical, cognitive and linguistic ability to carry out all aspects of the study

Exclusion Criteria:

* Reversible cause of HF (thyroid disorders, severe anemia, etc.)
* Hyponatremia at baseline (sodium <130 mmol/L)
* eGFR at baseline <30mL/min/1.73m2
* Scheduled cardiac surgery, coronary intervention (percutaneous coronary intervention or coronary artery bypass graft surgery) within 3 months
* Myocardial infarction within 3 months
* Comorbidity for which fluid restriction or unlimited fluid intake is advised
* Life expectancy <6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
B-lines | 12 weeks
  The patients will be investigated with lung ultrasound to screen for B-lines (comet tail artifacts) to assess pulmonary congestion
NT-proBNP | 12 weeks
  Specific biomarkers for heart failure (blood test)

SECONDARY OUTCOMES:
Heart failure symptoms | 12 weeks
  Symptoms of heart failure measured by questionnaires
HRQoL | 12 weeks
  Health related quality of life measured with EQ5D
Thirst distress | 12 weeks
Self-Care | 12 weeks
  Self-care in chronic illness, measured by a questionnaire
IVC | 12 weeks
  Ultrasound of Inferior Vena Cava (IVC) diameter and respiratory variation.
Pleural effusion | 12 weeks
  Lungultrasound with screening for pleural effusion
Physical Capacity | 12 weeks
  Physical Capacity measured by six minutes walktest
Hospital readmissions | 12 weeks
  Hospital readmissions within three months
Heart failure events | 12 weeks
  Contact with helathcare due to heart failure symtoms, increased use of diuretics with/without admission etc.

CONTACTS AND LOCATIONS:
Overall Officials: Carolin Nymark, PhD, Principal Investigator — Karolinska Universitetssjukhuset, Heart and Vascular Center
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No